CLINICAL TRIAL: NCT07180485
Title: The Effectiveness of Whole Body Vibration Training in Improving Brain Activity, Bone Mineral Density, Quality of Life, and Biomarkers for the Older People With Dynapenic Abdominal Obesity
Brief Title: Effectiveness of Whole Body Vibration on Health Outcomes in Older Adults With Dynapenic Abdominal Obesity
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dalin Tzu Chi General Hospital (Other)
Collaborators: Buddhist Dalin Tzu Chi General Hospital (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: B11401015; DTCRD113-E-14 (Other Grant/Funding Number: Buddhist Dalin Tzu Chi Hospital)
Record Dates: First submitted 2025-05-21; First posted 2025-09-18 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-05

CONDITIONS: Dynapenia; Abdominal Obesity
Keywords: whole-body vibration training; brain activity; bone mineral density; quality of life; biomarkers
MeSH Terms: conditions — Obesity, Abdominal | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- whole body vibration training group (Experimental): Participants in the experimental group underwent whole-body vibration (WBV) training three times per week for a total duration of 24 weeks. During each session, participants stood barefoot on a vibration platform, maintaining a static squat position with knees bent at 30 degrees and feet shoulder-width apart. The training protocol gradually increased in duration, number of sets, and total exercise time from an initial 10 minutes to 30 minutes over the 24-week period. The vibration frequency was progressively raised from 20 Hz to 40 Hz, with a constant amplitude of 2 mm. Each 10-minute session included a 1-minute rest interval. Additionally, all participants were provided with the "Move for Health" handbook issued by the Health Promotion Administration, Ministry of Health and Welfare, Taiwan, as part of health education guidance. Post-intervention data collection was conducted at weeks 18 and 25 following the 24-week intervention program.
  Interventions: Behavioral: whole body vibration training
- control group (Placebo Comparator): The control group received the "Move for Health" handbook issued by the Health Promotion Administration, Ministry of Health and Welfare, Taiwan, and participated in 30-minute health education sessions over a 24-week period. The educational content included exercise-related information, an introduction to dynapenic abdominal obesity (DAO), associated risk factors, and potential health consequences. Post-intervention data collection was conducted at weeks 18 and 25 following the 24-week intervention program.
  Interventions: Behavioral: control group

INTERVENTIONS:
Behavioral: whole body vibration training — whole body vibration training and health education booklet
  Arms: whole body vibration training group
Behavioral: control group — health education booklet
  Arms: control group

SUMMARY:
This study focuses on whole body vibration training (WBVT), a form of neuromuscular training that uses mechanical vibrations. WBVT has been shown to improve muscle function, bone mineral density, and quality of life. While some benefits have been observed in the elderly population, there remains a research gap concerning its effectiveness in older adults with dynapenic abdominal obesity. Therefore, the findings of this study will provide new evidence for health interventions targeting this specific group.

This research targets outpatients aged 65 and above who meet the criteria for dynapenic abdominal obesity. It aims to evaluate the effects of WBVT on brain activity, osteoporosis, quality of life, and biological markers. The study period is from February 1, 2025, to January 31, 2027, with a planned sample size of 120 participants, equally divided into an experimental group and a control group (60 participants each).

DETAILED DESCRIPTION:
The purpose of this study is to investigate the effects of whole body vibration training on older adults with dynapenic abdominal obesity in the following areas:

Brain activity: Changes in serum levels of brain-derived neurotrophic factor (BDNF).

Bone mineral density: Measured using dual-energy X-ray absorptiometry (DXA).

Quality of life: Assessed through questionnaires covering improvements in physical health, mental well-being, and social functioning.

Biomarkers: Changes in levels of total cholesterol, high- and low-density lipoprotein cholesterol, C-reactive protein (CRP), and glycated hemoglobin (HbA1c).

ELIGIBILITY:
Inclusion Criteria:

Outpatients aged 65 years or older

Diagnosed with dynapenic abdominal obesity

Able to understand and follow simple instructions

Able to communicate clearly and express their own will

Willing to sign the informed consent form

Exclusion Criteria:

Inability to communicate in Mandarin or Taiwanese, resulting in inability to participate in research activities

Severe visual or hearing impairment that hinders study participation

Presence of cognitive impairment, musculoskeletal or severe osteoporosis-related conditions

Refusal to sign the informed consent form

Ages: 65 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2027-10-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
blood tests | 24 weeks
  Total Cholesterol (TC) Time Frame: Baseline, 3 months, 6 months；Description: Serum total cholesterol level measured in mg/dL. Reference value: < 200 mg/dL.
  Triglycerides (TG) Time Frame: Baseline, 3 months, 6 months；Description: Serum triglyceride level measured in mg/dL. Reference value: < 150 mg/dL.
  Low-Density Lipoprotein Cholesterol (LDL-C) Time Frame: Baseline, 3 months, 6 months；Description: Serum LDL cholesterol measured in mg/dL. Reference value: < 130 mg/dL.
  High-Density Lipoprotein Cholesterol (HDL-C)Time Frame: Baseline, 3 months, 6 months；Description: Serum HDL cholesterol measured in mg/dL. Reference values: > 40 mg/dL for men, > 50 mg/dL for women.
  C-Reactive Protein (CRP)Time Frame: Baseline, 3months, 6 months；Description: Quantitative serum CRP level measured in mg/dL. Normal reference value: 0.3 mg/dL.
  Glycated Hemoglobin (HbA1c)Time Frame: Baseline, 3 months, 6 months；Description: HbA1c percentage measured in blood. Normal Brain-Derived Neurotroph in pg/mL using
dual-energy X-ray absorptiometry(DXA) | 8 months
  This study employed dual-energy X-ray absorptiometry (DXA), a widely used and clinically safe method for assessing bone health. The DXA system (brand referenced in previous publications) operates by emitting a low-radiation dose (±10 μSv) X-ray beam to measure the extent of X-ray penetration through body tissues. Based on the absorption data, the device calculates bone mineral density (BMD). Since bones absorb more X-rays and have high penetrability, while fat absorbs less and has low penetrability, DXA effectively differentiates between tissue types. DXA results are typically interpreted using T-scores for BMD. A T-score ≥ -1.0 indicates normal bone density and good skeletal health. A T-score between -2.5 and -1.0 suggests low bone mass (osteopenia), indicating a decreased BMD but not yet at the threshold for osteoporosis. A T-score ≤ -2.5 defines osteoporosis, indicating significantly reduced BMD and a higher risk of fractures. Severe osteoporosis is diagnosed when a T-score ≤ -2.5.
quality of life questionnaire | 24 weeks
  The Taiwan version of the World Health Organization Quality of Life questionnaire is a shortened version derived from the original 100-item WHOQOL-100 developed by the World Health Organization. Exploratory and confirmatory factor analyses of the questionnaire support a four-domain model consisting of physical health, psychological well-being, social relationships, and environment. The internal consistency (Cronbach's α) of these four domains ranges from 0.70 to 0.77. The questionnaire includes 28 items: one item for overall quality of life, one for general health, seven for physical health, six for psychological well-being, three for social relationships, and eight for environmental factors. The scale uses a 5-point Likert format based on frequency, intensity, capability, and evaluation. Higher scores indicate better quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Chang Shu Fang, professor, Study Chair — National Taipei University of Nursing and Health Sciences

IPD SHARING:
Plan to Share IPD: Yes
can sharing topics and research protocol
Supporting Information: Study Protocol
Time Frame: approximate date since June 2025 to January 2027
URL: https://orcid.org/0000-0002-8823-6901

REFERENCES:
- [Background] Zago M, Capodaglio P, Ferrario C, Tarabini M, Galli M. Whole-body vibration training in obese subjects: A systematic review. PLoS One. 2018 Sep 5;13(9):e0202866. doi: 10.1371/journal.pone.0202866. eCollection 2018. PMID 30183742
- [Background] Zhang L, Liu S, Wang W, Sun M, Tian H, Wei L, Wu Y. Dynapenic abdominal obesity and the effect on long-term gait speed and falls in older adults. Clin Nutr. 2022 Jan;41(1):91-96. doi: 10.1016/j.clnu.2021.11.011. Epub 2021 Nov 15. PMID 34864458
- [Background] Zhang J, Wang R, Zheng Y, Xu J, Wu Y, Wang X. Effect of Whole-Body Vibration Training on Muscle Activation for Individuals with Knee Osteoarthritis. Biomed Res Int. 2021 Mar 26;2021:6671390. doi: 10.1155/2021/6671390. eCollection 2021. PMID 33855078
- [Background] Yao G, Chung CW, Yu CF, Wang JD. Development and verification of validity and reliability of the WHOQOL-BREF Taiwan version. J Formos Med Assoc. 2002 May;101(5):342-51. PMID 12101852
- [Background] Wang X, Jiang J, Hu W, Hu Y, Qin LQ, Hao Y, Dong JY. Dynapenic Abdominal Obesity and Risk of Heart Disease among Middle-Aged and Older Adults: A Prospective Cohort Study. J Nutr Health Aging. 2023;27(9):752-758. doi: 10.1007/s12603-023-1975-0. PMID 37754215
- [Background] Wolf D, Ayon-Olivas M, Sendtner M. BDNF-Regulated Modulation of Striatal Circuits and Implications for Parkinson's Disease and Dystonia. Biomedicines. 2024 Aug 5;12(8):1761. doi: 10.3390/biomedicines12081761. PMID 39200225
- [Background] Wang W, Wang S, Lin W, Li X, Andersen LL, Wang Y. Efficacy of whole body vibration therapy on pain and functional ability in people with non-specific low back pain: a systematic review. BMC Complement Med Ther. 2020 May 27;20(1):158. doi: 10.1186/s12906-020-02948-x. PMID 32460819
- [Background] Wu S, Ning HT, Xiao SM, Hu MY, Wu XY, Deng HW, Feng H. Effects of vibration therapy on muscle mass, muscle strength and physical function in older adults with sarcopenia: a systematic review and meta-analysis. Eur Rev Aging Phys Act. 2020 Sep 17;17:14. doi: 10.1186/s11556-020-00247-5. eCollection 2020. PMID 32963629
- [Background] Wang Z, Zhang X, Sun M. The application of whole-body vibration training in knee osteoarthritis. Joint Bone Spine. 2022 Mar;89(2):105276. doi: 10.1016/j.jbspin.2021.105276. Epub 2021 Sep 15. PMID 34536625
- [Background] Wen J, Leng L, Hu M, Hou X, Huang J. Effects of whole-body vibration training on cognitive function: A systematic review. Front Hum Neurosci. 2023 Feb 9;17:854515. doi: 10.3389/fnhum.2023.854515. eCollection 2023. PMID 36845880
- [Background] Uchida S, Kamiya K, Hamazaki N, Nozaki K, Ichikawa T, Nakamura T, Yamashita M, Maekawa E, Reed JL, Yamaoka-Tojo M, Matsunaga A, Ako J. Prognostic utility of dynapenia in patients with cardiovascular disease. Clin Nutr. 2021 Apr;40(4):2210-2218. doi: 10.1016/j.clnu.2020.09.050. Epub 2020 Oct 13. PMID 33873266
- [Background] Torres-Costoso A, Lopez-Munoz P, Martinez-Vizcaino V, Alvarez-Bueno C, Cavero-Redondo I. Association Between Muscular Strength and Bone Health from Children to Young Adults: A Systematic Review and Meta-analysis. Sports Med. 2020 Jun;50(6):1163-1190. doi: 10.1007/s40279-020-01267-y. PMID 32060751
- [Background] Tuttle CSL, Thang LAN, Maier AB. Markers of inflammation and their association with muscle strength and mass: A systematic review and meta-analysis. Ageing Res Rev. 2020 Dec;64:101185. doi: 10.1016/j.arr.2020.101185. Epub 2020 Sep 26. PMID 32992047
- [Background] Tan TC, Guo YY, Ho DJ, Sanwari NAB, Quek PH, Tan RS, Yap FS, Yang M, Yeung MT. Reference Values, Determinants and Regression Equation for the Timed-Up and Go Test (TUG) in Healthy Asian Population Aged 21 to 85 Years. Int J Environ Res Public Health. 2023 May 3;20(9):5712. doi: 10.3390/ijerph20095712. PMID 37174230
- [Background] Teixeira IA, Coutinho ESF, Marinho V, Castro-Costa E, Deslandes AC. Prevalence of dynapenia and overlap with disability, depression, and executive dysfunction. Rev Saude Publica. 2023 Aug 4;57:43. doi: 10.11606/s1518-8787.2023057004580. eCollection 2023. PMID 37556665
- [Background] Schiro G, Iacono S, Ragonese P, Aridon P, Salemi G, Balistreri CR. A Brief Overview on BDNF-Trk Pathway in the Nervous System: A Potential Biomarker or Possible Target in Treatment of Multiple Sclerosis? Front Neurol. 2022 Jul 12;13:917527. doi: 10.3389/fneur.2022.917527. eCollection 2022. PMID 35911894
- [Background] Sun JY, Huang WJ, Hua Y, Qu Q, Cheng C, Liu HL, Kong XQ, Ma YX, Sun W. Trends in general and abdominal obesity in US adults: Evidence from the National Health and Nutrition Examination Survey (2001-2018). Front Public Health. 2022 Oct 6;10:925293. doi: 10.3389/fpubh.2022.925293. eCollection 2022. PMID 36276394
- [Background] Srisaphonphusitti L, Manimmanakorn N, Manimmanakorn A, Hamlin MJ. Effects of whole body vibration exercise combined with weighted vest in older adults: a randomized controlled trial. BMC Geriatr. 2022 Nov 28;22(1):911. doi: 10.1186/s12877-022-03593-4. PMID 36443661
- [Background] Sampaio RAC, Sewo Sampaio PY, Uchida MC, Arai H. Management of Dynapenia, Sarcopenia, and Frailty: The Role of Physical Exercise. J Aging Res. 2020 Jan 31;2020:8186769. doi: 10.1155/2020/8186769. eCollection 2020. No abstract available. PMID 32089882
- [Background] Shantakumari N, Ahmed M. Whole body vibration therapy and cognitive functions: a systematic review. AIMS Neurosci. 2023 May 18;10(2):130-143. doi: 10.3934/Neuroscience.2023010. eCollection 2023. PMID 37426779
- [Background] Remer F, Keilani M, Kull P, Crevenna R. Effects of whole-body vibration therapy on pain, functionality, postural stability, and proprioception in patients with subacute and chronic non-specific low back pain: a systematic review. Wien Med Wochenschr. 2025 Feb;175(1-2):20-40. doi: 10.1007/s10354-023-01026-4. Epub 2023 Nov 24. PMID 37999785
- [Background] Ribeiro VGC, Lacerda ACR, Santos JM, Coelho-Oliveira AC, Fonseca SF, Prates ACN, Flor J, Garcia BCC, Tossige-Gomes R, Leite HR, Fernandes JSC, Arrieiro AN, Sartorio A, Sanudo B, Sa-Caputo DC, Bernardo-Filho M, Figueiredo PHS, Costa HS, Lima VP, Cardoso RF, Bastone AC, Soares LA, Mendonca VA, Taiar R. Efficacy of Whole-Body Vibration Training on Brain-Derived Neurotrophic Factor, Clinical and Functional Outcomes, and Quality of Life in Women with Fibromyalgia Syndrome: A Randomized Controlled Trial. J Healthc Eng. 2021 Nov 30;2021:7593802. doi: 10.1155/2021/7593802. eCollection 2021. PMID 34900203
- [Background] Ramirez PC, de Oliveira DC, de Oliveira Maximo R, de Souza AF, Luiz MM, Delinocente MLB, Steptoe A, de Oliveira C, da Silva Alexandre T. Is dynapenic abdominal obesity a risk factor for cardiovascular mortality? A competing risk analysis. Age Ageing. 2023 Jan 8;52(1):afac301. doi: 10.1093/ageing/afac301. PMID 36626317
- [Background] Roongbenjawan N, Siriphorn A. Accuracy of modified 30-s chair-stand test for predicting falls in older adults. Ann Phys Rehabil Med. 2020 Jul;63(4):309-315. doi: 10.1016/j.rehab.2019.08.003. Epub 2019 Sep 11. PMID 31520784
- [Background] Rossi AP, Urbani S, Fantin F, Nori N, Brandimarte P, Martini A, Zoico E, Mazzali G, Babbanini A, Muollo V, Zamboni M. Worsening Disability and Hospitalization Risk in Sarcopenic Obese and Dynapenic Abdominal Obese: A 5.5 Years Follow-Up Study in Elderly Men and Women. Front Endocrinol (Lausanne). 2020 Jun 30;11:314. doi: 10.3389/fendo.2020.00314. eCollection 2020. PMID 32695067
- [Background] Paineiras-Domingos LL, Sa-Caputo DDC, Francisca-Santos A, Reis-Silva A, Carvalho-Lima RP, Neves MFT, Xavier VL, Quinart H, Boyer FC, Sartorio A, Taiar R, Bernardo-Filho M. Can whole body vibration exercises promote improvement on quality of life and on chronic pain level of metabolic syndrome patients? A pseudorandomized crossover study. J Appl Physiol (1985). 2020 Apr 1;128(4):934-940. doi: 10.1152/japplphysiol.00068.2019. Epub 2020 Feb 20. PMID 32078471
- [Background] Picca A, Coelho-Junior HJ, Calvani R, Marzetti E, Vetrano DL. Biomarkers shared by frailty and sarcopenia in older adults: A systematic review and meta-analysis. Ageing Res Rev. 2022 Jan;73:101530. doi: 10.1016/j.arr.2021.101530. Epub 2021 Nov 25. PMID 34839041
- [Background] de Oliveira RDJ, de Oliveira RG, de Oliveira LC, Santos-Filho SD, Sa-Caputo DC, Bernardo-Filho M. Effectiveness of whole-body vibration on bone mineral density in postmenopausal women: a systematic review and meta-analysis of randomized controlled trials. Osteoporos Int. 2023 Jan;34(1):29-52. doi: 10.1007/s00198-022-06556-y. Epub 2022 Oct 25. PMID 36282343
- [Background] Ofir O, Buch A, Rouach V, Goldsmith R, Stern N, Monsonego-Ornan E. Association between abdominal obesity and fragility fractures among elderly Israeli women. Aging Clin Exp Res. 2020 Aug;32(8):1459-1467. doi: 10.1007/s40520-019-01347-8. Epub 2019 Sep 14. PMID 31522392
- [Background] Odano I, Maeyatsu F, Asari M, Yamaguchi S, Miura T, Taki Y. Whole-body vibration exercise and training increase regional CBF in mild cognitive impairment with enhanced cognitive function. Ann Nucl Med. 2022 Jan;36(1):82-94. doi: 10.1007/s12149-021-01687-4. Epub 2021 Nov 11. PMID 34762232
- [Background] Ourry V, Gonneaud J, Landeau B, Moulinet I, Touron E, Dautricourt S, Le Du G, Mezenge F, Andre C, Bejanin A, Sherif S, Marchant NL, Paly L, Poisnel G, Vivien D, Chocat A, Quillard A, Ferrand Devouge E, de la Sayette V, Rauchs G, Arenaza-Urquijo EM, Chetelat G; Medit-Ageing Research Group. Association of quality of life with structural, functional and molecular brain imaging in community-dwelling older adults. Neuroimage. 2021 May 1;231:117819. doi: 10.1016/j.neuroimage.2021.117819. Epub 2021 Feb 5. PMID 33549750
- [Background] Nawrat-Szoltysik A, Sieradzka M, Nowacka-Chmielewska M, Piejko L, Duda J, Brachman A, Polak A. Effect of Whole-Body Vibration Training on Selected Intrinsic Risk Factors in Women Aged 60+ at Fall Risk: A Randomized Controlled Trial. Int J Environ Res Public Health. 2022 Dec 19;19(24):17066. doi: 10.3390/ijerph192417066. PMID 36554961
- [Background] Moreira-Marconi E, Teixeira-Silva Y, Meirelles AG, Melo-Oliveira MES, Santos ACG, Reis-Silva A, Paineiras-Domingos LL, Seixas A, Dionello CDF, Sa-Caputo DDC, Bernardo-Filho M. Inflammatory Biomarker Responses to Whole-Body Vibration in Subjects with Different Clinical Status: A Systematic Review. Int J Environ Res Public Health. 2022 Nov 11;19(22):14853. doi: 10.3390/ijerph192214853. PMID 36429572
- [Background] Montgomery G, McPhee J, Paasuke M, Sipila S, Maier AB, Hogrel JY, Degens H. Determinants of Performance in the Timed Up-and-Go and Six-Minute Walk Tests in Young and Old Healthy Adults. J Clin Med. 2020 May 21;9(5):1561. doi: 10.3390/jcm9051561. PMID 32455757
- [Background] Murawska-Cialowicz E, Wiatr M, Cialowicz M, Gomes de Assis G, Borowicz W, Rocha-Rodrigues S, Paprocka-Borowicz M, Marques A. BDNF Impact on Biological Markers of Depression-Role of Physical Exercise and Training. Int J Environ Res Public Health. 2021 Jul 15;18(14):7553. doi: 10.3390/ijerph18147553. PMID 34300001
- [Background] Mou X, He B, Zhang M, Zhu Y, Ou Y, Chen X. Causal influence of muscle weakness on cardiometabolic diseases and osteoporosis. Sci Rep. 2023 Nov 15;13(1):19974. doi: 10.1038/s41598-023-46837-y. PMID 37968290
- [Background] de Oliveira Maximo R, de Oliveira DC, Ramirez PC, Luiz MM, de Souza AF, Delinocente MLB, Steptoe A, de Oliveira C, da Silva Alexandre T. Dynapenia, abdominal obesity or both: which accelerates the gait speed decline most? Age Ageing. 2021 Sep 11;50(5):1616-1625. doi: 10.1093/ageing/afab093. PMID 34087934
- [Background] Maestroni L, Read P, Bishop C, Papadopoulos K, Suchomel TJ, Comfort P, Turner A. The Benefits of Strength Training on Musculoskeletal System Health: Practical Applications for Interdisciplinary Care. Sports Med. 2020 Aug;50(8):1431-1450. doi: 10.1007/s40279-020-01309-5. PMID 32564299
- [Background] Maximo RO, de Oliveira DC, Ramirez PC, Luiz MM, de Souza AF, Delinocente MLB, Steptoe A, de Oliveira C, Alexandre TDS. Combination of dynapenia and abdominal obesity affects long-term physical performance trajectories in older adults: sex differences. Am J Clin Nutr. 2022 May 1;115(5):1290-1299. doi: 10.1093/ajcn/nqac023. PMID 35102379
- [Background] Mayoral LP, Andrade GM, Mayoral EP, Huerta TH, Canseco SP, Rodal Canales FJ, Cabrera-Fuentes HA, Cruz MM, Perez Santiago AD, Alpuche JJ, Zenteno E, Ruiz HM, Cruz RM, Jeronimo JH, Perez-Campos E. Obesity subtypes, related biomarkers & heterogeneity. Indian J Med Res. 2020 Jan;151(1):11-21. doi: 10.4103/ijmr.IJMR_1768_17. PMID 32134010
- [Background] Perez-Campos Mayoral L, Matias-Cervantes CA, Perez-Campos E, Romero Diaz C, Laguna Barrios LA, Pina Canseco MDS, Martinez Cruz M, Perez-Campos Mayoral E, Solorzano Mata CJ, Rodal Canales FJ, Martinez Ruiz H, Hernandez-Huerta MT. Associations of Dynapenic Obesity and Sarcopenic Obesity with the Risk of Complications in COVID-19. Int J Mol Sci. 2022 Jul 27;23(15):8277. doi: 10.3390/ijms23158277. PMID 35955411
- [Background] Li W, Chen M, Chen F, Li Y, Zhong Y, Lu Y, Zhang K, Yang F. Vitamin D combined with whole-body vibration training for the treatment of osteo-sarcopenia: study protocol for a randomized controlled trial. Trials. 2024 Sep 30;25(1):638. doi: 10.1186/s13063-024-08498-8. PMID 39350307
- [Background] Liu IT, Lee WJ, Lin SY, Chang ST, Kao CL, Cheng YY. Therapeutic Effects of Exercise Training on Elderly Patients With Dementia: A Randomized Controlled Trial. Arch Phys Med Rehabil. 2020 May;101(5):762-769. doi: 10.1016/j.apmr.2020.01.012. Epub 2020 Feb 19. PMID 32084347
- [Background] Lu L, Mao L, Feng Y, Ainsworth BE, Liu Y, Chen N. Effects of different exercise training modes on muscle strength and physical performance in older people with sarcopenia: a systematic review and meta-analysis. BMC Geriatr. 2021 Dec 15;21(1):708. doi: 10.1186/s12877-021-02642-8. PMID 34911483
- [Background] Lee K, Lee JY, Kim YH. Low Grip Strength and Muscle Mass Increase the Prevalence of Osteopenia and Osteoporosis in Elderly Women. Healthcare (Basel). 2021 Apr 16;9(4):476. doi: 10.3390/healthcare9040476. PMID 33923692
- [Background] Liu P, Li Y, Xiao Y, Li D, Liu L, Ma Y, Zheng W. Effects of whole-body vibration training with different frequencies on the balance ability of the older adults: a network meta-analysis. Front Physiol. 2023 Apr 17;14:1153163. doi: 10.3389/fphys.2023.1153163. eCollection 2023. PMID 37123276
- [Background] Lee SC, Wu LC, Chiang SL, Lu LH, Chen CY, Lin CH, Ni CH, Lin CH. Validating the Capability for Measuring Age-Related Changes in Grip-Force Strength Using a Digital Hand-Held Dynamometer in Healthy Young and Elderly Adults. Biomed Res Int. 2020 Apr 20;2020:6936879. doi: 10.1155/2020/6936879. eCollection 2020. PMID 32382565
- [Background] Lin TH, Chang SF, Liao MT, Chen YH, Tsai HC. The relationships between physical function, nutrition, cognitive function, depression, and sleep quality for facility-dwelling older adults with dynapenia. BMC Geriatr. 2023 May 8;23(1):278. doi: 10.1186/s12877-023-03847-9. PMID 37158860
- [Background] Lv D, Shen S, Chen X. Association Between Dynapenic Abdominal Obesity and Fall Risk in Older Adults. Clin Interv Aging. 2022 Apr 7;17:439-445. doi: 10.2147/CIA.S347053. eCollection 2022. PMID 35418747
- [Background] LeBoff MS, Greenspan SL, Insogna KL, Lewiecki EM, Saag KG, Singer AJ, Siris ES. The clinician's guide to prevention and treatment of osteoporosis. Osteoporos Int. 2022 Oct;33(10):2049-2102. doi: 10.1007/s00198-021-05900-y. Epub 2022 Apr 28. PMID 35478046
- [Background] Lai Z, Lee S, Chen Y, Wang L. Comparison of whole-body vibration training and quadriceps strength training on physical function and neuromuscular function of individuals with knee osteoarthritis: A randomised clinical trial. J Exerc Sci Fit. 2021 Jul;19(3):150-157. doi: 10.1016/j.jesf.2021.01.003. Epub 2021 Feb 2. PMID 33680003
- [Background] Kao CY, Su YC, Chang SF. The Relationship between Dynapenic Abdominal Obesity and Fall: A Systematic Review and Meta-Analysis of 15,506 Middle to Older Adults. J Clin Med. 2023 Nov 23;12(23):7253. doi: 10.3390/jcm12237253. PMID 38068305
- [Background] Kobayashi K, Imagama S, Ando K, Nakashima H, Machino M, Morozumi M, Kanbara S, Ito S, Inoue T, Yamaguchi H, Ishiguro N, Hasegawa Y. Dynapenia and physical performance in community-dwelling elderly people in Japan. Nagoya J Med Sci. 2020 Aug;82(3):415-424. doi: 10.18999/nagjms.82.3.415. PMID 33132426
- [Background] Jawed Y, Beli E, March K, Kaleth A, Loghmani MT. Whole-Body Vibration Training Increases Stem/Progenitor Cell Circulation Levels and May Attenuate Inflammation. Mil Med. 2020 Jan 7;185(Suppl 1):404-412. doi: 10.1093/milmed/usz247. PMID 32074302
- [Background] Hatanaka S, Sasai H, Shida T, Osuka Y, Kojima N, Ohta T, Abe T, Yamashita M, Obuchi SP, Ishizaki T, Fujiwara Y, Awata S, Toba K; IRIDE Cohort Study investigators. Association between dynapenia and cognitive decline in community-dwelling older Japanese adults: The IRIDE Cohort Study. Geriatr Gerontol Int. 2024 Mar;24 Suppl 1:123-129. doi: 10.1111/ggi.14749. Epub 2023 Dec 20. PMID 38116709
- [Background] Harijanto C, Lim A, Vogrin S, Duque G. Does Whole-Body Vibration Training Have a Concurrent Effect on Bone and Muscle Health? A Systematic Review and Meta-Analysis. Gerontology. 2022;68(6):601-611. doi: 10.1159/000519511. Epub 2021 Nov 15. PMID 34781288
- [Background] Gomez-Campos R, Vidal-Espinoza R, Goncalves EM, Langer RD, Borges JH, Castelli-Correia de Campos LF, Urra-Albornoz C, Sulla Torres J, Cossio-Bolanos M. Accuracy in body composition scanning by adult half-body DXA scanning. Nutr Hosp. 2023 Apr 20;40(2):362-367. doi: 10.20960/nh.04416. PMID 36926940
- [Background] Grande G, Vetrano DL, Kalpouzos G, Welmer AK, Laukka EJ, Marseglia A, Fratiglioni L, Rizzuto D. Brain Changes and Fast Cognitive and Motor Decline in Older Adults. J Gerontol A Biol Sci Med Sci. 2023 Feb 24;78(2):326-332. doi: 10.1093/gerona/glac177. PMID 36037020
- [Background] Garabiles MR, Shen ZZ, Yang L, Chu Q, Hannam K, Hall BJ. Investigating the Physical and Mental Health Nexus: a Network Analysis of Depression, Cardiometabolic Health, Bone Mass, and Perceived Health Status Among Filipino Domestic Workers. Int J Behav Med. 2023 Apr;30(2):234-249. doi: 10.1007/s12529-022-10087-5. Epub 2022 May 16. PMID 35578098
- [Background] Gkastaris K, Goulis DG, Potoupnis M, Anastasilakis AD, Kapetanos G. Obesity, osteoporosis and bone metabolism. J Musculoskelet Neuronal Interact. 2020 Sep 1;20(3):372-381. PMID 32877973
- [Background] Fettrow T, Hupfeld K, Tays G, Clark DJ, Reuter-Lorenz PA, Seidler RD. Brain activity during walking in older adults: Implications for compensatory versus dysfunctional accounts. Neurobiol Aging. 2021 Sep;105:349-364. doi: 10.1016/j.neurobiolaging.2021.05.015. Epub 2021 May 31. PMID 34182403
- [Background] Eyileten C, Sharif L, Wicik Z, Jakubik D, Jarosz-Popek J, Soplinska A, Postula M, Czlonkowska A, Kaplon-Cieslicka A, Mirowska-Guzel D. The Relation of the Brain-Derived Neurotrophic Factor with MicroRNAs in Neurodegenerative Diseases and Ischemic Stroke. Mol Neurobiol. 2021 Jan;58(1):329-347. doi: 10.1007/s12035-020-02101-2. Epub 2020 Sep 17. PMID 32944919
- [Background] Eglseer D, Traxler M, Bauer S. Association between the Intake of Different Protein Sources and Obesity Coexisting with Low Handgrip Strength in Persons near Retirement Age. Nutrients. 2022 Nov 5;14(21):4684. doi: 10.3390/nu14214684. PMID 36364946
- [Background] Ding W, Zhang Y, Zhang L, Wang Z, Yu J, Ji H. Successful aging and environmental factors in older individuals in urban and rural areas: A cross-sectional study. Arch Gerontol Geriatr. 2020 Nov/Dec;91:104229. doi: 10.1016/j.archger.2020.104229. Epub 2020 Aug 14. PMID 32871304
- [Background] Dominguez-Munoz FJ, Villafaina S, Garcia-Gordillo MA, Hernandez-Mocholi MA, Collado-Mateo D, Adsuar JC, Gusi N. Effects of 8-Week Whole-Body Vibration Training on the HbA1c, Quality of Life, Physical Fitness, Body Composition and Foot Health Status in People with T2DM: A Double-Blinded Randomized Controlled Trial. Int J Environ Res Public Health. 2020 Feb 18;17(4):1317. doi: 10.3390/ijerph17041317. PMID 32085626
- [Background] Dowling L, Cuthbertson DJ, Walsh JS. Reduced muscle strength (dynapenia) in women with obesity confers a greater risk of falls and fractures in the UK Biobank. Obesity (Silver Spring). 2023 Feb;31(2):496-505. doi: 10.1002/oby.23609. Epub 2022 Dec 11. PMID 36504327
- [Background] Dieli-Conwright CM, Parmentier JH, Sami N, Lee K, Spicer D, Mack WJ, Sattler F, Mittelman SD. Adipose tissue inflammation in breast cancer survivors: effects of a 16-week combined aerobic and resistance exercise training intervention. Breast Cancer Res Treat. 2018 Feb;168(1):147-157. doi: 10.1007/s10549-017-4576-y. Epub 2017 Nov 22. PMID 29168064
- [Background] Dupont J, Vercauteren L, Amini N, Lapauw L, De Schaepdryver M, Poesen K, Dedeyne L, Verschueren S, Tournoy J, Koppo K, Gielen E. Are inflammatory markers associated with sarcopenia-related traits in older adults with sarcopenia? - A cross-sectional analysis of the ENHANce study. Exp Gerontol. 2023 Jul;178:112196. doi: 10.1016/j.exger.2023.112196. Epub 2023 May 16. PMID 37156446
- [Background] Delinocente MLB, Luiz MM, de Oliveira DC, de Souza AF, Ramirez PC, de Oliveira Maximo R, Soares NC, Steptoe A, de Oliveira C, da Silva Alexandre T. Are Serum 25-Hydroxyvitamin D Deficiency and Insufficiency Risk Factors for the Incidence of Dynapenia? Calcif Tissue Int. 2022 Dec;111(6):571-579. doi: 10.1007/s00223-022-01021-8. Epub 2022 Sep 15. PMID 36109388
- [Background] Dhawan D, Sharma S. Abdominal Obesity, Adipokines and Non-communicable Diseases. J Steroid Biochem Mol Biol. 2020 Oct;203:105737. doi: 10.1016/j.jsbmb.2020.105737. Epub 2020 Aug 18. PMID 32818561
- [Background] Corbianco S, Cavallini G, Baldereschi G, Carboncini MC, Fiamingo FL, Bongioanni P, Dini M. Whole body vibration and treadmill training in Parkinson's disease rehabilitation: effects on energy cost and recovery phases. Neurol Sci. 2018 Dec;39(12):2159-2168. doi: 10.1007/s10072-018-3566-0. Epub 2018 Sep 19. PMID 30229379
- [Background] Cezar NOC, Ansai JH, Oliveira MPB, da Silva DCP, Gomes WL, Barreiros BA, Langelli TCO, de Andrade LP. Feasibility of improving strength and functioning and decreasing the risk of falls in older adults with Alzheimer's dementia: a randomized controlled home-based exercise trial. Arch Gerontol Geriatr. 2021 Sep-Oct;96:104476. doi: 10.1016/j.archger.2021.104476. Epub 2021 Jul 4. PMID 34260986
- [Background] Carey JJ, Chih-Hsing Wu P, Bergin D. Risk assessment tools for osteoporosis and fractures in 2022. Best Pract Res Clin Rheumatol. 2022 Sep;36(3):101775. doi: 10.1016/j.berh.2022.101775. Epub 2022 Aug 29. PMID 36050210
- [Background] Cao V, Clark A, Aggarwal B. Obesity and Severity of Menopausal Symptoms: a Contemporary Review. Curr Diab Rep. 2023 Dec;23(12):361-370. doi: 10.1007/s11892-023-01528-w. Epub 2023 Nov 24. PMID 37999882
- [Background] Chen H, Yi YY, Zhang SB, Xu HW, Fang XY, Tao-Hu, Wu DS, Wang SJ. Sarcopenic obesity defined by visceral adiposity was associated with osteoporotic vertebral fracture. Arch Osteoporos. 2022 Mar 6;17(1):41. doi: 10.1007/s11657-022-01087-9. PMID 35249182
- [Background] Cariati I, Bonanni R, Pallone G, Romagnoli C, Rinaldi AM, Annino G, D'Arcangelo G, Tancredi V. Whole Body Vibration Improves Brain and Musculoskeletal Health by Modulating the Expression of Tissue-Specific Markers: FNDC5 as a Key Regulator of Vibration Adaptations. Int J Mol Sci. 2022 Sep 8;23(18):10388. doi: 10.3390/ijms231810388. PMID 36142305
- [Background] Cobos-Palacios L, Ruiz-Moreno MI, Vilches-Perez A, Vargas-Candela A, Munoz-Ubeda M, Benitez Porres J, Navarro-Sanz A, Lopez-Carmona MD, Sanz-Canovas J, Perez-Belmonte LM, Mancebo-Sevilla JJ, Gomez-Huelgas R, Bernal-Lopez MR. Metabolically healthy obesity: Inflammatory biomarkers and adipokines in elderly population. PLoS One. 2022 Jun 9;17(6):e0265362. doi: 10.1371/journal.pone.0265362. eCollection 2022. PMID 35679338
- [Background] Chittrakul J, Siviroj P, Sungkarat S, Sapbamrer R. Multi-System Physical Exercise Intervention for Fall Prevention and Quality of Life in Pre-Frail Older Adults: A Randomized Controlled Trial. Int J Environ Res Public Health. 2020 Apr 29;17(9):3102. doi: 10.3390/ijerph17093102. PMID 32365613
- [Background] Califf RM. Biomarker definitions and their applications. Exp Biol Med (Maywood). 2018 Feb;243(3):213-221. doi: 10.1177/1535370217750088. PMID 29405771
- [Background] Carvalho AF, Maes M, Solmi M, Brunoni AR, Lange S, Husain MI, Kurdyak P, Rehm J, Koyanagi A. Is dynapenia associated with the onset and persistence of depressive and anxiety symptoms among older adults? Findings from the Irish longitudinal study on ageing. Aging Ment Health. 2021 Mar;25(3):468-475. doi: 10.1080/13607863.2019.1699021. Epub 2019 Dec 12. PMID 31829040
- [Background] Correa HL, Rosa TDS, Dutra MT, Sales MM, Noll M, Deus LA, Reis AL, de Araujo TB, Neves RVP, Gadelha AB. Association between dynapenic abdominal obesity and inflammatory profile in diabetic older community-dwelling patients with end-stage renal disease. Exp Gerontol. 2021 Apr;146:111243. doi: 10.1016/j.exger.2021.111243. Epub 2021 Jan 15. PMID 33460716
- [Background] Batsis JA, Zbehlik AJ, Pidgeon D, Bartels SJ. Dynapenic obesity and the effect on long-term physical function and quality of life: data from the osteoarthritis initiative. BMC Geriatr. 2015 Oct 8;15:118. doi: 10.1186/s12877-015-0118-9. PMID 26449277
- [Background] Bordoni A, Boesch C, Malpuech-Brugere C, Orfila C, Tomas-Cobos L. The role of bioactives in energy metabolism and metabolic syndrome. Proc Nutr Soc. 2019 Aug;78(3):340-350. doi: 10.1017/S0029665119000545. Epub 2019 Apr 10. PMID 30967168
- [Background] Bourdel-Marchasson I, Ostan R, Regueme SC, Pinto A, Pryen F, Charrouf Z, d'Alessio P, Baudron CR, Guerville F, Durrieu J, Donini LM, Franceschi C, Valentini L. Quality of Life: Psychological Symptoms-Effects of a 2-Month Healthy Diet and Nutraceutical Intervention; A Randomized, Open-Label Intervention Trial (RISTOMED). Nutrients. 2020 Mar 18;12(3):800. doi: 10.3390/nu12030800. PMID 32197408
- [Background] Beaumont M, Losq A, Peran L, Berriet AC, Couturaud F, Le Ber C, Reychler G. Comparison of 3-minute Step Test (3MStepT) and 6-minute Walk Test (6MWT) in Patients with COPD. COPD. 2019 Aug;16(3-4):266-271. doi: 10.1080/15412555.2019.1656713. Epub 2019 Sep 5. PMID 31581920
- [Background] Bragg AE, Crowe-White KM, Ellis AC, Studer M, Phillips F, Samsel S, Parton J, Locher JL, Ard JD. Changes in Cardiometabolic Risk Among Older Adults with Obesity: An Ancillary Analysis of a Randomized Controlled Trial Investigating Exercise Plus Weight Maintenance and Exercise Plus Intentional Weight Loss by Caloric Restriction. J Acad Nutr Diet. 2022 Feb;122(2):354-362. doi: 10.1016/j.jand.2021.07.009. Epub 2021 Sep 1. PMID 34486528
- [Background] Burt LA, Billington EO, Rose MS, Raymond DA, Hanley DA, Boyd SK. Effect of High-Dose Vitamin D Supplementation on Volumetric Bone Density and Bone Strength: A Randomized Clinical Trial. JAMA. 2019 Aug 27;322(8):736-745. doi: 10.1001/jama.2019.11889. PMID 31454046
- [Background] Bemben D, Stark C, Taiar R, Bernardo-Filho M. Relevance of Whole-Body Vibration Exercises on Muscle Strength/Power and Bone of Elderly Individuals. Dose Response. 2018 Dec 6;16(4):1559325818813066. doi: 10.1177/1559325818813066. eCollection 2018 Oct-Dec. PMID 30559636
- [Background] Ali N, Mohanto NC, Nurunnabi SM, Haque T, Islam F. Prevalence and risk factors of general and abdominal obesity and hypertension in rural and urban residents in Bangladesh: a cross-sectional study. BMC Public Health. 2022 Sep 8;22(1):1707. doi: 10.1186/s12889-022-14087-8. PMID 36076233
- [Background] da Silva Alexandre T, Scholes S, Ferreira Santos JL, de Oliveira Duarte YA, de Oliveira C. Dynapenic Abdominal Obesity Increases Mortality Risk among English and Brazilian Older Adults: A 10-Year Follow-Up of the ELSA and SABE Studies. J Nutr Health Aging. 2018;22(1):138-144. doi: 10.1007/s12603-017-0966-4. PMID 29300433
- [Background] Ahmad A, Imran M, Ahsan H. Biomarkers as Biomedical Bioindicators: Approaches and Techniques for the Detection, Analysis, and Validation of Novel Biomarkers of Diseases. Pharmaceutics. 2023 May 31;15(6):1630. doi: 10.3390/pharmaceutics15061630. PMID 37376078
- [Background] Afshar PF, Wiig EH, Malakouti SK, Shariati B, Nejati S. Reliability and validity of a quick test of cognitive speed (AQT) in screening for mild cognitive impairment and dementia. BMC Geriatr. 2021 Dec 15;21(1):693. doi: 10.1186/s12877-021-02621-z. PMID 34911461
- [Background] Ayan G, Afacan C, Poyraz BC, Bilgic O, Avci S, Yavuzer H, Yuruyen M, Erdincler DS, Ayan B, Doventas A. Reliability and Validity of Rowland Universal Dementia Assessment Scale in Turkish Population. Am J Alzheimers Dis Other Demen. 2019 Feb;34(1):34-40. doi: 10.1177/1533317518802449. Epub 2018 Oct 17. PMID 30328357
- See also: Related Info — https://orcid.org/0000-0002-8823-6901
- Available data/document: Study Protocol: t780927t@yahoo.com.tw — https://orcid.org/0000-0002-8823-6901 — t780927t@yahoo.com.tw